CLINICAL TRIAL: NCT05597904
Title: Genetic and Biological Background and Follow-up of Different Phenotypes of Coeliac Disease
Brief Title: Background of Different Phenotypes of Coeliac Disease
Status: Recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other); University of Turku (Other); Oulu University Hospital (Other); University of Debrecen (Other); University of Trieste (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Teea Salmi, Professor in Dermatology, Tampere University Hospital
Other Study IDs: R22088
Record Dates: First submitted 2022-10-03; First posted 2022-10-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Celiac Disease; Dermatitis Herpetiformis
Keywords: coeliac disease; dermatitis herpetiformis; gluten-free diet; transglutaminase; microbiata
MeSH Terms: conditions — Celiac Disease; Dermatitis Herpetiformis | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Coeliac disease patients: Adult (18 years or over) patients with previous coeliac disease or dermatitis herpetiformis diagnosis
  Interventions: Genetic: Genetic predisposition
- Healthy controls: 500 adult (18 years or over) friends or non-related family members of coeliac disease or dermatitis herpetiformis patients participating in the study, no previous coeliac disease or dermatitis herpetiformis diagnosis. In addition 1000 controls will be included from Biobank
  Interventions: Genetic: Genetic predisposition

INTERVENTIONS:
Genetic: Genetic predisposition — Assessment of genetic predisposition to various celiac disease phenotypes. No intervention.

SUMMARY:
The main purpose of this study is to investigate genetic, serological, immunological and microbiata diversities between different coeliac disease phenotypes and to discover applicable prognostic markers for specific phenotypes.

DETAILED DESCRIPTION:
The recognition of clinical heterogeneity has expanded the understanding of coeliac disease, but the factors contributing to this diversity remain unclear. Moreover, since coeliac disease is highly heterogeneous, there is a need for more individualized follow-up and support and implementation of more personalized follow-up guidelines.

In this study coeliac disease and dermatitis herpetiformis patients and healthy controls will be recruited. Genetic, clinical, immunological, micobiata and novel biomedical markers are compared between coeliac disease phenotypes and also controls and their prognostic value is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Cohorts 1 and 2: coeliac disease or dermatitis herpetiformis diagnosis
* Cohort 3: friend or non-related family member of coeliac disease or dermatitis herpetiformis patient

Exclusion Criteria:

* Cohorts 1-3: Age <18 years
* Cohorts 1 and 2: coeliac disease or dermatitis herpetiformis diagnosis not confirmed
* Cohort 3: coeliac disease or dermatitis herpetiformis diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: National and also focused recruitment for patients with coeliac disease or dermatitis herpetiformis diagnosis. Healthy controls recruited via volunteered subjects with coeliac disease or dermatitis herpetiformis
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-HLA variant association | baseline
  phenotype specific non-HLA variants

SECONDARY OUTCOMES:
serum transglutaminase antibodies | baseline
  Levels of serum antibodies against transglutaminase
microbiata | baseline
  skin and intestinal microbiata findings
quality of life measure | baseline
  PGWB questionnaire (22-items with values 1-6, total score range 22-132, a higher score indicating better quality of life)
gastrointestinal symptoms | baseline
  GSRS-questionnaire (15 items with values 1-7, total score 1-7 as a mean value of all scores, higher score indicating more severe symptoms)
dietary adherence | baseline
  strictness of gluten-free diet (GIP-test)

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No